CLINICAL TRIAL: NCT03149250
Title: Characteristics of Primary and Plasmatic Hemostasis in Preeclampsia - a Cross-sectional Study
Brief Title: Characteristics of Primary and Plasmatic Hemostasis in Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Christian F. Weber, MD, Prof. Dr. med. Christian F. Weber, Cooperative Weichteilsarkom Study Group
Other Study IDs: Hemostasis_Preeclampsia
Record Dates: First submitted 2017-05-03; First posted 2017-05-11 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Coagulation Disorder, Blood; Platelet Function
Keywords: Aggregometry
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant Preeclampsia: Pregnant between 35th and 40th week of pregnancy Preeclampisa
  Intervention: Aggregometry, Monitoring of plasmatic hemostasis: Aggregometry and conventional coagulation testing after blood sampling in the context of routinely performed blood sampling
  Interventions: Diagnostic Test: Aggregometry, Monitoring of plasmatic hemostasis
- Pregnant No-Preeclampsia: Control Group 1 Pregnant between 35th and 40th week of pregnancy No Preeclampsia Healthy Intervention: Aggregometry, Monitoring of plasmatic hemostasis: Aggregometry and conventional coagulation testing after blood sampling in the context of routinely performed blood sampling
  Interventions: Diagnostic Test: Aggregometry, Monitoring of plasmatic hemostasis
- Not Pregnant: Control group 2 Healthy and not pregnant control group
  Intervention: Aggregometry, Monitoring of plasmatic hemostasis: Aggregometry and conventional coagulation testing after blood sampling.
  Interventions: Diagnostic Test: Aggregometry, Monitoring of plasmatic hemostasis

INTERVENTIONS:
Diagnostic Test: Aggregometry, Monitoring of plasmatic hemostasis — Multiple Electrode Aggregometry using the Multiplate system Coagulation factor analyses (FXIII, FVIII, vWF) Parameters of conventional coagulation testing (aPTT, INR, Platelet count)

SUMMARY:
The study aims to investigate the impact of preeclampsia on hemostasis.

DETAILED DESCRIPTION:
In comparison to healthy pregnant women and non-pregnant woman, this study analyses parameters of primary hemostasis and plasmatic coaguation in preeclamptic pregnant woman. Detailed analyses of the platelet function is performed using the Multiple Electrode Aggregometry, detailed analyses of the plasmatic coagulation syste is performed by isolated coaguation factor analyses and conventional coagulation analyses.

ELIGIBILITY:
Inclusion Criteria:

* Platelet count > 100 / nll
* In study group and control group 1: Week of Pregnancy: 35-40
* in control group 2: healthy, not pregnant woman

Exclusion Criteria:

* Hereditary coagulopathy
* Missing content of the patient / proband
* Eclampsia
* HELLP syndrome
* CRP > 1 mg/dl
* Fever (> 38°C)

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female (Study cohort is pregnant, control group should be female too)
Study Population: Pregnant patients suffering from preeclampsia, n = 20
  Control group 1: Healthy pregnant patients, not suffering from preeclampsia, n=20
  Control group 2: Healthy woman (age between 18 and 40y) that are not pregnant
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Area under the aggregation curve in the ADPtest of the Multiple Electrode Aggregometry | Between 35th and 40th week of pregnancy; in control group 2 (not pregnant) within 1 week after inclusion into the study
  ADP induced platelet aggregation

SECONDARY OUTCOMES:
Area under the aggregation curve in the ASPItest of the Multiple Electrode Aggregometry | Between 35th and 40th week of pregnancy; in control group 2 (not pregnant) within 1 week after inclusion into the study
  Arachidonic acid induced platelet aggregation
Area under the aggregation curve in the TRAPtest of the Multiple Electrode Aggregometry | Between 35th and 40th week of pregnancy; in control group 2 (not pregnant) within 1 week after inclusion into the study
  Thrombin induced platelet aggregation
Parameters of plasmatic coagulation system | Between 35th and 40th week of pregnancy; in control group 2 (not pregnant) within 1 week after inclusion into the study
  von Willebrand Factor, Factor VIII, Factor XIII, parameter of conventional coagulation testing (apTT, INR, platelet count, Fibrinogen)

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, MD, PhD, Principal Investigator — Goethe University

IPD SHARING:
Plan to Share IPD: No